CLINICAL TRIAL: NCT02809248
Title: The Influence Cirrhosis of the Liver on the Coronary Re-stenosis (LTX-Stent Study)
Brief Title: The Influence Cirrhosis of the Liver on the Coronary Re-stenosis (LTX- Stent Study)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the small number of patients, none could be included in the study.
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-123
Record Dates: First submitted 2016-06-06; First posted 2016-06-22 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Re-stenosis; Cirrhosis of the Liver
Keywords: LTX Study
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- coated stent (Active Comparator): the patient get a coated coronary stent implantation (ZES - zotarolimus eluting stent)
  Interventions: Device: ZES
- uncoated stent (Active Comparator): the patient get a uncoated coronary stent implantation (BMS - bare metal stent)
  Interventions: Device: BMS

INTERVENTIONS:
Device: ZES — stent implantation (zotarolimus eluting stent)
  Arms: coated stent
Device: BMS — stent implantation (bare metal stent)
  Arms: uncoated stent

SUMMARY:
The aim of the study is to choose an optimal stent and to get further knowledge about the mechanisms of the engraftment of a stent.

The occurrence of a hyperplasia of neointima can be minimized by application of a coated stent and a concurrent safety four weekly dual thrombocytes therapy

ELIGIBILITY:
Inclusion Criteria:

* male and female patients with a severe dysfunction of liver
* patient is planned a coronary stent implantation
* adults who are contractually capable and mentally able to understand and follow the instructions of the study personnel
* written informed consent prior to study participation

Exclusion Criteria:

* younger than 18 years
* pregnancy and breast-feeding
* acute cardiac syndrome
* contraindication against an intracardiac catheter
* persons in dependence from the sponsor or working with the sponsor
* participation in a parallel interventional clinical trial
* patient has been committed to an institution by legal or regulatory order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2017-12 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
the ideal stent (coated stent or uncoated stent) | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Becker, MD, Principal Investigator — Uniklinik RWTH Aachen, Med. Klinik I

IPD SHARING:
Plan to Share IPD: No